CLINICAL TRIAL: NCT04565093
Title: Efficacy of iPACK (Interspace Between the Popliteal Artery and the Capsule of the Posterior Knee) Versus Periarticular Local Infiltration Analgesia After Unilateral Total Knee Arthroplasty: Prospective Randomized Control Trial
Brief Title: Efficacy of iPACK After Unilateral TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University Hospital (Other)
Responsible Party: Principal Investigator, Abdul Sattar Narejo, Consultant Anesthesiologist, King Khalid University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB PROJECT NO. E-20-4819
Record Dates: First submitted 2020-09-11; First posted 2020-09-25 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Arthroplasty Complications; Pain, Joint; Arthritis Knee; Regional Anesthesia Morbidity
Keywords: Knee arthroplasty; Pain control; iPACK; Local infiltration analgesia; Early rehabilitation
MeSH Terms: conditions — Arthralgia; Agnosia

STUDY DESIGN:
Intervention Model Description: This study is conducted to evaluate posterior knee pain after unilateral Total Knee Arthroplasty (TKA) comparing iPACK (Interspace between the popliteal artery and the capsule of the posterior knee) and Periarticular Local Infiltration Analgesia (LIA) under spinal anesthesia. All patients will receive Adductor Canal Block (ACB) to cover pain from anteromedial aspect of knee. 169 adult patients will be recruited in this study and will be divided into two groups; group-1 iPACK (n=85) will receive Adductor Canal Block (ACB) + iPACK and group 2 LIA (n=84) will receive ACB+ periarticular Local Infiltration Analgesia (LIA). The primary outcome, severity of pain (NRS) will be evaluated in Post Anesthesia Care Unit (PACU). The secondary outcome, time to mobilization (ROM and TUG tests) along with pain score will be recorded in the ward after 2 hours of surgery then every 12 hours until the patient discharged home.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The data will be collected by the care provider (nurses & assistant anesthetists) and outcome assessors (physiotherapists) who will be unaware of group allocation and will record their findings in the patient's file and on a predesigned form. Patient's demographic data, duration of surgery, tourniquet time, PACU stay, postoperative heart rate, mean arterial pressure, pain score, knee range of motion (ROM), time-up-go (TUG), time to hospital discharge, patient and surgeon satisfaction, and any complication will be recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPACK (Experimental): In this group, participants will receive a peripheral nerve anesthetic block that is iPACK (Interspace between the Popliteal Artery and the Capsule of the posterior Knee) to cover posterior knee pain after total knee arthroplasty (TKA). This anesthetic block will be performed by assigned anesthesiologist under ultrasound guidance.
  Interventions: Procedure: iPACK
- Periarticular local infiltration analgesia (LIA) (Placebo Comparator): In this group, participants will receive a mixture of bupivacaine 0.25% 20 ml + epinephrine 100 mics ± lornoxicam 8 mg ± morphine 10 mg ± tranexamic acid 1 gm in 40 ml normal saline (NS) that will be injected into the posterior capsule and the medial and lateral ligaments just before implantation: after insertion of the implants and into the capsule and retinacular tissues. The remaining solution (approximately 20 mL) will be used to infiltrate the muscle and subcutaneous tissues. This local anesthetic infiltration is commonly performed by the operating orthopedic surgeon during TKA for postoperative pain control.
  Interventions: Procedure: Periarticular local infiltration analgesia (LIA)

INTERVENTIONS:
Procedure: iPACK — Interspace between the popliteal artery and the capsule of the posterior knee (iPACK):
  This is basically ultrasound guided peripheral nerve block performed by the anesthesiologists at the posterior side of the knee to control pain after TKA.
  Arms: iPACK
Procedure: Periarticular local infiltration analgesia (LIA) — A mixture of Bupivacaine 0.25% 20 ml + epinephrine 100 mics ± lornoxicam 8 mg ± morphine 10 mg ± tranexamic acid 1 gm in 40 ml normal saline (NS) will be injected into the posterior capsule and the medial and lateral ligaments just before implantation: after insertion of the implants and into the capsule and retinacular tissues. The remaining solution (approximately 20 mL) will be used to infiltrate the muscle and subcutaneous tissues. This intervention is commonly performed by the operating orthopedic surgeon to control pain after TKA.
  Arms: Periarticular local infiltration analgesia (LIA)

SUMMARY:
Total knee arthroplasty (TKA) is a common orthopedic procedure associated with severe postoperative pain which may limit patient rehabilitation and hospital discharge. Although various analgesic techniques have been proposed, there is currently no consensus on the optimal protocol to improve functional outcomes following TKA. The ideal analgesic regimen post TKA should enable adequate pain control, early mobilization and physical therapy, shorten hospital stay, reduce the risk of postoperative complications and improve patient satisfaction. Our hypothesis is iPACK (Interspace between the Popliteal Artery and the Capsule of the posterior Knee) peripheral nerves anesthetic block is superior to Periarticular local Infiltration Analgesia (LIA)which is commonly given by the surgeons during the TKA in terms of pain relief and early mobilization.

DETAILED DESCRIPTION:
Background: Total Knee Arthroplasty (TKA) is one of the most frequent procedures performed by orthopedic surgeons. Research has found that orthopedic surgeries are the most painful procedures.(1) Unrelieved pain post orthopedic surgery is a stressor that can cause altered physiologic changes and negative effects on every organ system of the body. Untreated pain can result in complex pathophysiology than the pain caused by the original injury or disease. This can have both detrimental physical and psychological consequences for patients, as well as a substantial economic impact due to increased costs of health care and lost productivity. (2) The anatomy of sensory supply to the knee joint is complex with contributions from both the lumbar and sacral plexuses. The anterior-medial compartmental innervation consists of branches from the femoral nerve, including the saphenous nerve, the medial femoral cutaneous nerve and the nerve to vastus medialis. The lateral femoral cutaneous nerve, the common peroneal nerve, and the nerves to vastus intermedius and lateralis innervate the knee anterolaterally. The posterior group consists of the popliteal nerve plexus that ramifies around the genicular vasculature in the popliteal fossa. The popliteal nerve plexus is derived from the tibial nerve and the posterior branch of the obturator nerve. The posterior group supplies intra-articular innervation to the menisci, the peri-meniscular joint capsule, the cruciate ligaments, the infra-patellar fat pad, and the posterior part of the fibrous knee capsule.(3) The medial para-patellar arthrotomy performed for total knee arthroplasty, through the anteromedial integument of the knee and the extra-articular medial retinacular complex, evokes pain mediated by the infra-patellar branch of the saphenous nerve, the medial retinacular nerve (the terminal branch of the nerve to vastus medialis), and the anterior branch of the medial femoral cutaneous nerve. This procedure will not affect the extra-articular nerve branches to the anterolateral portion of the knee from the common peroneal nerve, the nerves to vastus intermedius and lateralis, and the lateral femoral cutaneous nerve. The intra-articular excision evokes pain from structures innervated by the posterior group. (4) Ultrasound-guided Femoral Nerve Block (FNB) is one of the most commonly used techniques that has been shown to significantly improve analgesia and reduce postoperative opioid consumption after TKA. However, FNB may lead to quadriceps muscle weakness, limiting ambulation and increasing the risk of falls, making physical rehabilitation results unsatisfactory.(5) Recently, there has been increased interest in the Adductor Canal Block (ACB) for pain relief after total knee arthroplasty. (6) The adductor canal is a pyramidal, musculoaponeurotic tunnel from the apex of the femoral triangle to the adductor hiatus, running between the vastus medialis muscle anterolaterally and the adductor longus and adductor Magnus muscles posteromedially. It is covered in its entire length by the vastoadductor membrane. The contents of the adductor canal include the superficial artery and vein, saphenous nerve, the nerve to vastus medialis, the posterior branch of the obturator nerve, and in some cases, the medial cutaneous nerve and the anterior branch of the obturator nerve. The advantage of this technique rests in the fact that it provides localized motor-sparing analgesia, with similar opioid consumption and side effects when compared with FNB.(7) However, ACB does not provide analgesia to the posterior aspect of the knee, which can be moderate to severe after surgery. This pain may be ameliorated by the addition of the ultrasound-guided local anesthetic infiltration of the Interspace between the Popliteal Artery and the Capsule of the posterior Knee (iPACK). (8) Although this technique seems to provide many advantages, it may present some limitations and risks like intravascular injection and injury due to the presence of the popliteal vessels near the target. Although the use of ultrasound guidance decreases this risk, significant bleeding and serious complications can still occur due to the inability to recognize and compress the source of bleeding. (4)

Methods: In this study we are going to recruit 169 participants to compare them in two groups. group-1 iPACK (n=85) will receive Adductor Canal Block (ACB) + iPACK and group 2 LIA (n=84) ACB+ periarticular Local Infiltration Analgesia (LIA). All participants, care provider (nurses & assistant anesthetists) and outcome assessors (physiotherapist) will be blinded to the group allocation. Only the anesthesiologist responsible for perioperative care performing the ACB and iPACK blocks will be aware of the randomization. All peripheral nerve blocks will be performed with complete aseptic technique and under ultrasound guidance. Periarticular LIA will be performed by the surgeon with the landmark technique base. This study will be conducted in six months' duration. All patients will consent for spinal anesthesia, ACB, and iPACK and they will be instructed how to report pain on a 10 cm long Numerical Rating Scale (NRS) postoperatively.

The primary outcome, severity of pain (NRS) will be evaluated in Post Anesthesia Care Unit (PACU). The secondary outcome, time to mobilization along with pain score will be recorded in the ward after 2 hours of surgery then every 12 hours until the patient discharged home. Quadriceps muscle strength will be evaluated with the knee range of motion (ROM). A completely straight knee joint (extension) will measure 0° and a fully bent knee will have a flexion of at 130° degrees. The Timed-Up-and-Go (TUG) tests to evaluate functional recovery after TKA. The TUG test measures the time it takes a patient to get up from a chair, walk 3 m, and return to the sitting position in the chair.

On arrival to operation room (OR), all eligible participants will have intravenous (IV) cannula in situ and monitors according to the Association of Anesthetists of Great Britain and Ireland (AAGBI). Under complete aseptic technique, spinal anesthesia will be performed with pencil point 25 Gauge (Whitacre) needle with heavy Bupivacaine 0.5% and Fentanyl 15 micrograms (mics) total 3 milliliters (ml). After spinal anesthesia, each participant will receive either ultrasound-guided ACB+iPACK or ACB+ periarticular LIA.

Description of peripheral nerve blocks technique:

Adductor Canal Block (ACB): The skin is disinfected and the transducer (SonoSite 8-14 MHz) is placed anteromedially, approximately at the junction between the middle and distal third of the thigh. The saphenous nerve is usually identified as anterior and lateral to the femoral artery. The needle (Pajunk Germany100 mm) will be inserted in-plane from lateral-to-medial orientation and advanced toward the femoral artery deep to the sartorius muscle. Once the needle tip is visualized anterior to the artery and after careful aspiration, 1-2 mL of local anesthetic will be injected to confirm the proper injection site. If injection of local anesthetic does not appear to result in its spread around the femoral artery, additional needle repositions and injections may be necessary. A total of 20 millilitres (ml) of Bupivacaine 0.25% will be injected.

Interspace between the popliteal artery and the capsule of the posterior knee (iPACK):

The patient will be placed in a supine position with the lower extremity flexed at the knee and abducted at the hip. To begin scanning, the transducer will be placed on the lower third of the medial thigh to visualize the femur and the femoral vessels in cross-section. The transducer then will be slide caudally to observe the femoral artery as it dives into the popliteal fossa through the adductor hiatus to become the popliteal artery. At this point, the transducer will be moved posteriorly and inferiorly to visualize the space between the popliteal artery and the shaft of the femur just superior to the femoral condyles. The needle will be inserted, in a plane, from the anterior end of the transducer in a medial to the lateral trajectory, keeping the needle parallel to the acoustic shadow of the femur. With the needle tip resting 2 cm beyond the lateral border of the artery, 20 mL of Bupivacaine 0.25% will be injected, after negative aspiration of blood, to infiltrate the tissue space in divided doses as the needle is withdrawn.

Periarticular Local Infiltration Analgesia (LIA):

A mixture of Bupivacaine 0.25% 20 ml + epinephrine 100 mics ± lornoxicam 8 mg ± morphine 10 mg ± tranexamic acid 1 gm in 40 ml normal saline (NS) will be injected into the posterior capsule and the medial and lateral ligaments just before implantation: after insertion of the implants and into the capsule and retinacular tissues. The remaining solution (approximately 20 mL) will be used to infiltrate the muscle and subcutaneous tissues.

Postoperatively all participants will be prescribed 1 gm Paracetamol oral every 6 hours + buprenorphine transdermal patch 5 mics ± celecoxib 200 mg every 12 hours ± oxycodone 10 mg every 12 hours ± pregabalin 75 mg every 12 hours for breakthrough pain.

Sample Size:

In King Khalid University Hospital, we are approximately doing annually 300 TKA cases. Assuming that and confidence level of 95%, margin of error 5% Raosoft® recommended sample size is 169.

Data Collection:

The data will be collected by the outcome assessors who will be unaware of group allocation and will record their findings in patient's file and on predesigned form. Patients demographic data, duration of surgery, tourniquet time, PACU stay, postoperative heart rate, mean arterial pressure, pain score, knee range of motion (ROM), time-up-go (TUG), time to hospital discharge, patient and surgeon satisfaction and any complication will be recorded.

Statistical Analysis:

Statistical analysis was performed using Statistical Package for the Social Sciences (SPSS) version 24.0 software (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status score I-III
* Scheduled for elective unilateral TKA
* Age > 18 < 80 years
* BMI < 40 kg/m2

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status score (ASA) IV
* Patient scheduled for revision of TKA
* Rheumatoid Arthritis patient
* Prior back surgery
* Patients on any anticoagulant
* Any other contra-indication for spinal anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-27 (Actual)

PRIMARY OUTCOMES:
Change from preoperative pain score after TKA | Through study completion, an average of 3 days
  The pain will assessed by numerical rating scale (NRS). From 0 to 10, with 0 being no pain and 10 being the worst pain imaginable

SECONDARY OUTCOMES:
Knee range of motion (ROM) | Through study completion, an average of 3 days
  The functional recovery of the knee joint after TKA will be evaluated by ROM.A completely straight knee joint (extension) will measure 0° and a fully bent knee will have a flexion of at 130° degrees
Timed-up and go (TUG) | Through study completion, an average of 3 days
  The functional recovery of the knee joint after TKA will be evaluated by TUG test. The TUG test is the time it takes a patient to get up from a chair, walk 3 m, and return to the sitting position in the chair

OTHER OUTCOMES:
Any other adverse event related to peripheral nerve blocks | Through study completion, an average of 3 days
  Any injury related to nerve blocks like Common Peroneal Nerve Block (CPN) or injury, Vascular injury, Compartment syndrome, Myositis, local anesthesia systemic toxicity (LAST), prolong anesthetic block

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Sattar Narejo, FCPS, FCAI, Principal Investigator — King Saud University College of Medicine and King Khalid University Hospital
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results
Supporting Information: Study Protocol, SAP
Time Frame: The IPD will be available starting from January 2022 to December 2022
Access Criteria: The IPD study protocol and statistical analysis will be accessible on request by email to the principal investigator.

REFERENCES:
- [Result] YaDeau JT, Cahill JB, Zawadsky MW, Sharrock NE, Bottner F, Morelli CM, Kahn RL, Sculco TP. The effects of femoral nerve blockade in conjunction with epidural analgesia after total knee arthroplasty. Anesth Analg. 2005 Sep;101(3):891-895. doi: 10.1213/01.ANE.0000159150.79908.21. PMID 16116010
- [Result] Fine PG. Long-term consequences of chronic pain: mounting evidence for pain as a neurological disease and parallels with other chronic disease states. Pain Med. 2011 Jul;12(7):996-1004. doi: 10.1111/j.1526-4637.2011.01187.x. PMID 21752179
- [Result] Runge C, Borglum J, Jensen JM, Kobborg T, Pedersen A, Sandberg J, Mikkelsen LR, Vase M, Bendtsen TF. The Analgesic Effect of Obturator Nerve Block Added to a Femoral Triangle Block After Total Knee Arthroplasty: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):445-51. doi: 10.1097/AAP.0000000000000406. PMID 27171822
- [Result] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Result] Jiang X, Wang QQ, Wu CA, Tian W. Analgesic Efficacy of Adductor Canal Block in Total Knee Arthroplasty: A Meta-analysis and Systematic Review. Orthop Surg. 2016 Aug;8(3):294-300. doi: 10.1111/os.12268. PMID 27627711
- [Result] Grevstad U, Mathiesen O, Valentiner LS, Jaeger P, Hilsted KL, Dahl JB. Effect of adductor canal block versus femoral nerve block on quadriceps strength, mobilization, and pain after total knee arthroplasty: a randomized, blinded study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):3-10. doi: 10.1097/AAP.0000000000000169. PMID 25376972
- [Result] Thobhani S, Scalercio L, Elliott CE, Nossaman BD, Thomas LC, Yuratich D, Bland K, Osteen K, Patterson ME. Novel Regional Techniques for Total Knee Arthroplasty Promote Reduced Hospital Length of Stay: An Analysis of 106 Patients. Ochsner J. 2017 Fall;17(3):233-238. PMID 29026354
- See also: King Khalid University Hospital — https://medicalcity.ksu.edu.sa/en/page/king-khalid-university-hospital